CLINICAL TRIAL: NCT00004049
Title: A Phase I and Pharmacokinetic Study of SR-45023A Administered Once Every 7 Days
Brief Title: SR-45023A in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: CDR0000067233; ILEX-SR102-A4; SACI-IDD-99-06; NCI-V99-1560
Record Dates: First submitted 1999-12-10; First posted 2004-05-03 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2001-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — apomine

INTERVENTIONS:
Drug: apomine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of SR-45023A in treating patients who have locally advanced or metastatic solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of SR-45023A in patients with locally advanced or metastatic solid tumors. II. Determine the quantitative and qualitative toxic effects of SR-45023A in these patients. III. Assess the plasma and urine pharmacokinetics of SR-45023A and relate these to drug effects, if possible, in these patients. IV. Determine any preliminary antitumor activity of SR-45023A in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral SR-45023A weekly. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SR-45023A until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed for up to 1 month.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced or metastatic solid tumors refractory to standard therapy or for which no standard therapy exists (surgery, radiotherapy, and/or chemotherapy) Measurable or evaluable disease by medical photograph, plain x-ray, CT, MRI, palpation, or serum tumor markers at least 2 times upper limit of normal No symptomatic, progressive brain metastases by CT or MRI scan No cerebral edema No leukemia or multiple myeloma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL No coagulation disorders Hepatic: Bilirubin normal AST and ALT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver involvement) PT or INR, and PTT normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No cardiac conduction abnormalities Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active or uncontrolled infection No other concurrent severe disease No known hypersensitivity to SR-45023A analogs No concurrent or recent (within past 6 months) small bowel obstruction, symptoms of small bowel obstruction, or any other gastrointestinal disease impacting absorption of study drug No psychiatric disorders or geographic distance that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks since carboplatin, mitomycin, or nitrosoureas) and recovered No prior SR-45023A No other concurrent chemotherapy Endocrine therapy: No concurrent steroid therapy for brain disease No concurrent hormonal cancer therapy (except contraception, hormone replacement therapy, or corticosteroids) Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy (except symptomatic radiotherapy for pathologic fractures) Surgery: At least 4 weeks since prior surgery and recovered Other: At least 4 weeks since prior investigational agents No other concurrent investigational agents No concurrent anticoagulation therapy (e.g., heparin) except low dose warfarin for central venous catheter patency No concurrent digoxin, beta blockers, or calcium channel blockers No concurrent H2 histamine inhibitors (e.g., ranitidine, famotidine, or cimetidine), proton pump inhibitors (e.g., omeprazole or lansoprazole), or other drugs that might interfere with study drug absorption

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Drug Development, San Antonio, Texas, United States